CLINICAL TRIAL: NCT05104047
Title: Moxibustion for Neuropathic Pain in Type 2 DM
Brief Title: Distal Peripheral Neuropathy in Type 2 Diabetes
Acronym: DSP/DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S17-00829
Record Dates: First submitted 2021-10-16; First posted 2021-11-02 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Neuropathy; Pain, Neuropathic; Diabetes
Keywords: neuropathy, pain, neuropathic pain, diabetes, moxibustion
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia; Diabetes Mellitus; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional Moxibustion (Active Comparator): Participants receive Active Traditional Moxibustion - a protocol aimed at reducing neuropathic pain/discomfort.
  Interventions: Other: Moxibustion - Traditional (Active)
- Smokeless Moxibustion (Active Comparator): Participants receive Active Smokeless Moxibustion - a protocol aimed at reducing neuropathic pain/discomfort.
  Interventions: Other: Moxibustion - Smokeless - (Active)
- Placebo Moxibustion Control (Placebo Comparator): Participants receive Placebo Moxibustion - a protocol that mimics the active protocol but is not.
  Note. All participants randomized to the Control will be offered active protocol moxibustion treatments, at no cost, at the end of their study participation.
  Interventions: Other: Placebo Moxibustion
- Waitlist Control (No Intervention): WaitList (Control) No treatment. Subjects receive all aspects of study participation with the exception of exposure to Moxibustion.
  Note. All participants randomized to the Control will be offered active protocol moxibustion treatments, at no cost, at the end of their study participation.

INTERVENTIONS:
Other: Moxibustion - Traditional (Active) — Traditional Moxibustion (Moxa) is a technique in which the herb, artemisia, in a cigar shape (pole moxa) is lit (burned) and applied over specific acupuncture points which follows a specific protocol aimed at reducing neuropathic lower limb pain/discomfort.
  Other Names: Moxa (abreviation)
  Arms: Traditional Moxibustion
Other: Moxibustion - Smokeless - (Active) — Smokeless Moxibustion uses the same technique as traditional moxa however, the moxa is smokeless. Smokeless moxa allows for use in a broad range of treatment settings. The protocol is aimed at reducing neuropathic lower limb pain/discomfort.
  Other Names: Moxa (abreviation)
  Arms: Smokeless Moxibustion
Other: Placebo Moxibustion — Participants receive Placebo Moxibustion - a protocol that mimics the active protocol but is not active.
  Arms: Placebo Moxibustion Control

SUMMARY:
Distal sensory peripheral neuropathy (DSP) is a chronic, debilitating painful condition affecting quality of life in persons living with Type 2 diabetes. Treatments prescribed to manage DSP pain, such as nonnarcotic and narcotic analgesics, antidepressants and anticonvulsants, are largely ineffective. This is a preliminary study at assessing the feasibility, efficiency and preliminary efficacy of a novel non-pharmacologic pain management approach, moxibustion, to reduce DSP pain and improve quality of life.

DETAILED DESCRIPTION:
Distal sensory peripheral neuropathy (DSP) is a chronic, debilitating painful condition affecting quality of life in persons with Type 2 diabetes mellitus (T2DM). According to the Centers for Disease Control (CDC), 29 million Americans are living with T2DM. Treatments prescribed to manage DSP pain, such as nonnarcotic and narcotic analgesics, antidepressants and anticonvulsants, are largely ineffective. Effective management of DSP pain is an unmet therapeutic need for this population.

This is a randomized, blinded, placebo-controlled clinical trial to determine feasibility and preliminary efficacy of Moxibustion (Moxa) for persons with T2DM DSP lower limb pain/discomfort. Participants with lower limb DSP pain/discomfort are randomized to one of four Conditions: 1) Traditional Moxa, 2) Smokeless Moxa 3) Placebo Moxa (control), or 4) WaitList (control). Participation involves a preliminary phone screening, provider verification of medical condition, intake baseline session, neurologicial evaluations, treatment sessions and follow ups. Participants assigned to the moxibustion conditions will be blind to treatment assignment, attend a screening session, followed by twice-weekly treatment sessions for 3 weeks, complete the same instruments and submit prospective symptom diaries (SD). Subjects randomized to the WaitList control condition experience all aspects of study participation with the exception of receiving moxibustion (during the study). They undergo all screening and eligibility assessments; attend study visits; submit and review their symptom diaries, update concomitant medication, complete assessment instruments; receive neuro/NST assessments and compensation. In all respects, participants in the Control groups receive the same concern as subjects assigned to the other groups. All moxibustion interventions will be implemented by licensed acupuncturists.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-75 years of age, with a history of chronic bilateral neuropathic foot pain (pain, numbness, tingling) secondary to T2DM for the past three months or greater.
* Gracely Pain Scale (GPS) rated pain severity at "moderate" or above, documented in 1-week prospective self report symptom diary (SD)(a).
* Primary care provider (PCP) verification of T2DM diagnosis, report of neuropathic foot pain.
* Successfully complete a mini-mental status exam (obtaining a score of 24 or above).
* Must understand and agree to complete daily symptom diaries for the duration of the study.
* If on pharmacologic treatment(s) must have 21 days of stable regimen (same drugs, dose & frequency) prior to enrollment.

Exclusion Criteria:

* Any acute condition requiring medical care (severe heart disease, uncontrolled hypertension, lung disease, renal failure, foot lesions, sores, ingrown nails, infection etc.).
* Use topically applied medications to the lower extremities / feet.
* Allergic to smoke
* Alcohol and/or substance dependence.
* Receiving injectable corticosteroids.
* Receiving other complementary therapies such as herbs, massage, acupuncture etc. for foot pain.
* Pregnant women.
* Relocation or other plans that interfere with attending all of the planned study session and/or recording SD information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Gracely Pain Scale | Change from baseline rating of pain/discomfort (Gracely Pain Scale) after 3 wks of twice-wkly treatment sessions (the end of the treatment phase)
  The GPS is a Likert magnitude-estimation log-scale of sensory pain. Subjects rate their DSP pain by selecting one of 13 words to describe their average and worst DSP pain.
  "Nothing"=0 to "Extremely intense"=12

SECONDARY OUTCOMES:
Subjective Peripheral Neuropathy Screen (SPNS) | Change from baseline rating of neuropathy symptoms after 3 wks of twice-wkly treatment sessions (the end of the treatment phase)
  Describes neuropathy symptoms eg. aching/burning, "pins and needles", numbness, location (hands/arms, feet/legs), and severity of symptoms from "minimal" to "extreme".

OTHER OUTCOMES:
Clinical Global Severity & Improvement Scale | Change from baseline rating of pain intensity after 3 wks of twice-wkly treatment sessions (the end of the treatment phase)
  The severity of illness scale measures global severity of symptoms [in the context of peripheral neuropathy]. The patient rates discomfort from peripheral neuropathy on a scale of 0= No discomfort to 6= Very severe discomfort. The global improvement component measures the level of change from initial severity: 0= No improvement at all to 6= Great improvement
Neurological Sensory Testing (NST) | Change from baseline neurological physical assessment after 3 wks of twice-wkly treatment sessions
  Neurological assessments with Neuro Sensory Testing (NST) include: muscle strength and reflexes and sensory testing for lower limb vibration, pain and thermal sensation. Standard neurological assessment: muscle strength 0-5; reflexes 0-5; pain- intact, reduced, absent, hyperalgesia; vibration - intact, impaired; thermal - intact, reduced absent. The neuro/NST also serves to monitor for clinical safety and findings

CONTACTS AND LOCATIONS:
Overall Officials: J. Anastasi, PhD, Principal Investigator — New York University
Locations (2):
- United States (2):
  - New York University, Division of Special Studies in Symptom Management, New York, New York
  - NYU Special Studies in Symptom Management, New York, New York

IPD SHARING:
Plan to Share IPD: No